CLINICAL TRIAL: NCT01928043
Title: Adjunctive Curcumin for Symptomatic Adolescents With Bipolar Disorder: Brain and Body Considerations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: The Depressive and Bipolar Disorder Alternative Treatment Foundation (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Associate Professor, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 443-2011
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- adjunctive curcumin (Experimental): Curcumin will be added to their current medications for 8 weeks. Starting dose will be 500mg daily, increased to 500mg twice daily in week 2, then increased to 1000mg twice daily during weeks 3-8. A slower titration will be used for subjects who demonstrate tolerability problems.
  Interventions: Drug: Curcumin

INTERVENTIONS:
Drug: Curcumin
  Other Names: turmeric

SUMMARY:
This study will enroll 30 adolescents with bipolar disorder (BD) who are suffering from symptoms of depression despite already taking a traditional mood-stabilizing medication. Curcumin will be added to their current medications for 8 weeks. During these 8 weeks, their mood symptoms will be assessed regularly. Height, weight, and blood pressure will also be measured repeatedly. Blood tests will be completed before treatment, after 4 weeks of treatment, and at the end of the study. Blood tests will allow us to determine whether changes in inflammation and oxidative stress explain curcumin's effect on mood. Finally, we will use sophisticated technology to measure blood vessel functioning. We have three main predictions: 1. Curcumin will improve mood symptoms without causing physical problems; 2. Curcumin will reduce inflammation and oxidative stress, and these reductions will be linked to improvements in mood; 3. Curcumin will improve blood vessel functioning, and these improvements will be linked to improved inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* all races and ethnicities
* bipolar disorder I or II
* currently treated with lithium, divalproex, lamotrigine, and/or second generation antipsychotic
* doses stable for greater than or equal to 4 weeks
* current CGI BP score of moderate or greater
* current CDRS-R severity of greater than or equal to 35

Exclusion Criteria:

* If female, pregnant or sexually active without reliable contraception
* significant suicidal ideations (as determined by clinical interview or CDRS-R > 3) and/or any suicidal intent, even if fleeting or non-recurrent, in the preceding 2 weeks
* substance dependence within the past 2 months
* daily antidepressant, glucocorticoid, nonsteroidal anti-inflammatory, anti-platelet, anti-coagulant, antacid, or oral hypoglycemic medication or insulin; high-dose antioxidant vitamin supplements or other natural health products that may function as an antidepressant within 30 days of baseline
* IQ<80 or autistic disorder
* full threshold mania and/or YMRS > 20 and/or psychosis
* hypersensitivity to curcumin/turmeric, gelatin
* dietary consumption of curcumin/turmeric > 3 times/week
* clinically significant or unstable medical disorder; known gallstones and/or bile duct obstruction, stomach ulcers, excessive stomach acid/heartburn/gastroesophageal reflux disease (GERD); or clinically significant baseline laboratory abnormalities; or ALT and /or AST above the upper limit of normal on repeat examination at baseline
* severe depression (CDRS-R > 98) and/or severely ill (CGI BP >5)

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2013-09; Primary Completion 2017-03-03 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale - Revise (CDRS-R) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Measures mood symptom severity. Response is defined as greater than or equal to 50% reduction in CDRS-R score.
Oxidative Stress Markers | Change from baseline to endpoint (measured at weeks 0, 4, 8)
  Obtained through blood work
Pro-Inflammatory Markers | Change from baseline to endpoint (measured at weeks 0, 4, 8)
  Obtained through blood work
Endothelial Function | Change from baseline to endpoint (measured at weeks 0, 4, 8)
  Will be assessed via RH-PAT using the EndoPAT

SECONDARY OUTCOMES:
Clinical Global Impression - Bipolar Disorder Version (CGI BP) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Measures overall illness severity. Remission is defined as an improvement score of 1 or 2.
KSADS Depression Section (KDRS) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Measures mood symptoms severity
KSADS Mania Rating Scale (KMRS) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Measures symptoms severity
Young Mania Rating Scale (YMRS) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Measures symptom severity
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Change from baseline to endpoint (assessed at weeks 0, 2, 4, 6, 8)
  Anxiety self-report
Weight Gain | Change from baseline to endpoint (measured at 0, 4, 8)
  Significant weight gain is greater than or equal to 7% of baseline weight
Blood Pressure | Change from baseline to endpoint (measured at 0, 4, 8)
Side Effects for Children and Adolescents (SEFCA) | Change from baseline to endpoint (assessed at weeks 0, 4, 6, 8)
  SEFCA is a questionnaire that assesses side effects. We anticipate that no major side-effects will have a prevalence of greater than 20%.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada